CLINICAL TRIAL: NCT06663254
Title: Safety and Efficacy of Perioperative Volume Replacement with Volulyte 6% in Moderate-to-high Cardiovascular Risk Patients Having Major Abdominal Surgery: a Parallel-group, Double-blind Randomized Trial
Brief Title: Safety and Efficacy of Perioperative Volume Replacement with Volulyte 6% in Moderate-to-high Cardiovascular Risk Patients Having Major Abdominal Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XiangyaHMZKHES; 2024060725 (Other: Xiangya Hospital Medical Ethics Committee)
Record Dates: First submitted 2024-09-05; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Perioperative Volume Replacement; Hydroxyethyl Starch
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Specifically, everyone except anesthesia clinicians will be blinded to treatment. Anesthesia clinicians who are not blinded will conduct treatment and record intraoperative conditions. Outcome assessors responsible for postoperative follow-up are blinded to patient randomization; Statistical analysis performed independently by the designated blinded statistician. Emergency unblinding will only be done by an investigator and/or dedicated authorized personnel (e.g., the Pharmacovigilance Department of the Sponsor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6% hydroxyethyl starch 130/0.4 (Experimental)
  Interventions: Drug: Hydroxyethyl starch 130/0.4
- Sodium acetate Ringer (Other)
  Interventions: Drug: Sodium acetate Ringer

INTERVENTIONS:
Drug: Hydroxyethyl starch 130/0.4 — Individualized goal-directed administration of 6% Hydroxyethyl starch (HES) 130/0.4: After the induction of anesthesia, 200 ml trial fluid will be infused over 20 min. If stroke volume (SV) increases >10%, another 200 ml fluid will be given. After that, the use of trial fluid will be determined by the patients' Stroke Volume Variation (SVV). If the SVV exceeds 12%, 200 ml trial fluid will be given over 20 min; this will be repeated until SVV <12%. If the use of HES exceeds 30 ml/kg, sodium acetate Ringer will be replaced. In addition, patients will have a background infusion of sodium acetate Ringer's solution at 4 ml/kg/h to satisfy the maintenance fluid requirements during surgery.
  Other Names: Volulyte 6%; 6% Hydroxyethyl starch 130/0.4
  Arms: 6% hydroxyethyl starch 130/0.4
Drug: Sodium acetate Ringer — Individualized goal-directed administration of crystalloid alone: After the induction of anesthesia, 200 ml trial fluid will be infused over 20 min.
  If stroke volume (SV) increases >10%, another 200 ml fluid will be given. After that, the use of trial fluid will be determined by the patients' Stroke Volume Variation (SVV). If the SVV exceeds 12%, 200 ml trial fluid will be given over 20 min; this will be repeated until SVV <12%. In addition, patients will have a background infusion of sodium acetate, the maintenance fluid requirement during surgery.
  Arms: Sodium acetate Ringer

SUMMARY:
The investigators propose a multicenter randomized trial to test the renal safety of 6% hydroxyethyl starch (HES) 130/0.4 combined with sodium acetate Ringer's crystalloid solution in moderate-to-high cardiovascular risk patients having major abdominal surgery. The reference group will only be given sodium acetate Ringer's crystalloid.

DETAILED DESCRIPTION:
The investigators propose a multicenter randomized trial to test the renal safety of 6% hydroxyethyl starch (HES) 130/0.4 combined with sodium acetate Ringer's crystalloid solution in moderate-to-high cardiovascular risk patients having major abdominal surgery. The reference group will only be given sodium acetate Ringer's crystalloid.

The investigators will test the primary hypothesis that the maximum decrease in serum Cystatin-C-based estimated glomerular filtration rate (eGFR) from preoperatively through the initial 3 postoperative hospital days is non-inferior in patients who are randomized to a goal-directed combination of HES and crystalloid volume replacement versus goal-directed crystalloid alone.

Secondarily, the investigators will determine the long-term renal safety (cystatin C-based eGFR on postoperative 1 and 3 months) of HES and its effect on major adverse cardiovascular events and the length of hospitalization. Exploratory outcomes will include intraoperative hemodynamic indices, postoperative gastrointestinal indicators, the rate of unscheduled transferring to intensive care unit, the incidence of hospital re-admission within 30 days, the incidence of renal replacement therapy within 90 days after surgery, and the incidence of acute kidney injury based on serum creatine within 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 45 years old;
* Scheduled for elective open or laparoscopic gastrointestinal surgery expected to last ≥2 hours;
* Having general anesthesia;
* Expected to require at least overnight hospitalization;
* Subject to at least one of the following risk factors:

  1. Age ≥65 years;
  2. History of peripheral arterial disease;
  3. History of coronary artery disease;
  4. History of stroke or transient ischemic attack;
  5. Diabetes requiring medication;
  6. Current smoking or 15-pack-year history of smoking tobacco;
  7. Body mass index ≥30 kg/m2;
  8. Preoperative high-sensitivity troponin T ≥14 ng/L or troponin I equivalent, defined as ≥15 ng/L (Abbott assay), 19 ng/L (Siemens assay), or 25% of the 99% percentile for other assays - all within 6 months;
  9. B-type natriuretic protein (BNP) ≥80 ng/L or N-terminal B-type natriuretic protein (NT-ProBNP) ≥200 ng/L within six months.

Exclusion Criteria:

* Participate in conflicting studies;
* Are designated American Society of Anesthesiologists physical status 4;
* Are pregnant and/or breastfeeding;
* Have hypoproteinemia (serum albumin <30 g/L) or were given preoperative intravenous colloids, including albumin;
* Have recent intracranial or cerebral hemorrhage;
* Have preoperative acute kidney injury or chronic renal insufficiency (Serum Creatine ≥140 µmol/L for men, Serum Creatine≥120 µmol/L for women and/or oliguria/anuria) or renal replacement therapy;
* Have severe hepatic impairment (Alanine Transaminase (ALT) and/or Aspartate Aminotransferase (AST) more than two times the upper limit of normal);
* Are in congestive heart failure or have pulmonary edema;
* Are critically ill or septic;
* Have electrolyte disorders such as hypernatremia, hyperchloremia, hyperkalemia, or severe alkalosis;
* Are fluid overloaded or dehydrated;
* Have clinically meaningful coagulation or bleeding disorders;
* Had a solid organ transplant;
* Have a current serious burn injury;
* Have a mental illness that precludes adequate consent or cooperation with the proposed trial;
* Have known hypersensitivity or contraindication to Volulyte 6% or any sodium acetate Ringer solution component.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Maximum change in serum Cystatin-C based estimated glomerular filtration rate (eGFR) from baseline through initial 3 postoperative hospital days | Baseline and postoperative 1/2/3 day
  The decrease in cystatin-C-based eGFR from preoperatively to the minimum value recorded during the initial three postoperative hospital days. Increases in postoperative eGFR will be considered a reduction of 0 for analysis purposes.

SECONDARY OUTCOMES:
Cystatin-C based eGFR on postoperative 1 month | Postoperative 1 month
  The absolute value of cystatin-C based eGFR on postoperative 1 month.
Cystatin-C based eGFR on postoperative 3 months | Postoperative 3 months
  The absolute value of cystatin-C based eGFR on postoperative 3 months.
Postoperative major adverse cardiovascular events composite | Postoperative 30 days
  Major adverse cardiovascular events are a composite of all-cause mortality or one or more of the following cardiovascular complications occurring within 30 days after surgery: myocardial injury after non-cardiac surgery (MINS), non-fatal cardiac arrest, stroke, ventricular arrhythmia requiring treatment.
The length of hospitalization | Postoperative 3 month

OTHER OUTCOMES:
Average cardiac index | Perioperative
Responses to boluses of each fluid | Perioperative
  The average difference between the cardiac index measured before a bolus is given and of the cardiac index measured 30 after the beginning of each bolus.
Total fluid volume | Perioperative and the subsequent first 24 postoperative hours
  Total fluid volume (sodium Acetate Ringer and 6% hydroxyethyl starch 130/0.4) given during anesthesia and the subsequent first 24 postoperative hours.
Generalized average real variability of mean arterial pressure | Perioperative
Time to first defecation | Postoperative 30 days
Time to tolerance of oral liquid diet | Postoperative 30 days
Postoperative gastrointestinal complications | Postoperative 30 days
  Postoperative gastrointestinal complications occurring by day 30 after surgery (defined as the need for surgical reoperation): anastomotic leakage, leakage of the rectum, intestinal obstruction, peritonitis, necrosis of stoma, et, at. which need reoperation or endoscopic drainage.
Hospital re-admission within 30 days | Postoperative 30 days
The rate of unscheduled transferring to intensive care unit (ICU) | Postoperative 30 days
the incidence of acute kidney injury based on available serum creatine | Postoperative 7 days
The incidence of renal replacement therapy within 90 days after surgery | Postoperative 3 month

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of Zhengzhou University;, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shanxi
  - Chaoyang Hospital of Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for individual participant data meta-analysis.

REFERENCES:
- [Background] Reiterer C, Kabon B, Taschner A, Zotti O, Kurz A, Fleischmann E. A comparison of intraoperative goal-directed intravenous administration of crystalloid versus colloid solutions on the postoperative maximum N-terminal pro brain natriuretic peptide in patients undergoing moderate- to high-risk noncardiac surgery. BMC Anesthesiol. 2020 Aug 4;20(1):192. doi: 10.1186/s12871-020-01104-9. PMID 32753064
- [Background] Yates DR, Davies SJ, Milner HE, Wilson RJ. Crystalloid or colloid for goal-directed fluid therapy in colorectal surgery. Br J Anaesth. 2014 Feb;112(2):281-9. doi: 10.1093/bja/aet307. Epub 2013 Sep 20. PMID 24056586
- [Background] Futier E, Garot M, Godet T, Biais M, Verzilli D, Ouattara A, Huet O, Lescot T, Lebuffe G, Dewitte A, Cadic A, Restoux A, Asehnoune K, Paugam-Burtz C, Cuvillon P, Faucher M, Vaisse C, El Amine Y, Beloeil H, Leone M, Noll E, Piriou V, Lasocki S, Bazin JE, Pereira B, Jaber S; FLASH Trial Group; Lasocki S, Huet O, Cadic A, Jacob C, Paugam-Burtz C, Restoux A, Ouattara A, Feitita I, Deloge E, Defaye M, Joannes-Boyau O, Carles P, Napolitano G, Monziols S, Futier E, Vignaud M, Paul S, Gahbiche K, Fayon J, Laroche E, Bazin JE, Brandely A, Le Moal C, Lebuffe G, Garot M, Piriou V, Jaber S, Chanques G, Verzilli D, De Jong A, Millot A, Castagnoli A, Leone M, Pastene B, Castelli C, Medam S, Velly L, Vaisse C, Faucher M, Asehnoune K, Samba E, Roquilly A, Le Penndu M, Cuvillon P, Yves Lefrant J, Wira O, Dubout E, Mfam WS, Lescot T, Begneu E, Burey J, Cirilovic T, Beloeil H, Allo G, Pottecher J, Lebas B, Venot C, Rameau JP, Dimache F, Leger PS, El Amine Y. Effect of Hydroxyethyl Starch vs Saline for Volume Replacement Therapy on Death or Postoperative Complications Among High-Risk Patients Undergoing Major Abdominal Surgery: The FLASH Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):225-236. doi: 10.1001/jama.2019.20833. PMID 31961418
- [Background] Kabon B, Sessler DI, Kurz A; Crystalloid-Colloid Study Team. Effect of Intraoperative Goal-directed Balanced Crystalloid versus Colloid Administration on Major Postoperative Morbidity: A Randomized Trial. Anesthesiology. 2019 May;130(5):728-744. doi: 10.1097/ALN.0000000000002601. PMID 30882476
- [Background] Joosten A, Delaporte A, Ickx B, Touihri K, Stany I, Barvais L, Van Obbergh L, Loi P, Rinehart J, Cannesson M, Van der Linden P. Crystalloid versus Colloid for Intraoperative Goal-directed Fluid Therapy Using a Closed-loop System: A Randomized, Double-blinded, Controlled Trial in Major Abdominal Surgery. Anesthesiology. 2018 Jan;128(1):55-66. doi: 10.1097/ALN.0000000000001936. PMID 29068831
- [Background] Reiterer C, Kabon B, Halvorson S, Sessler DI, Mascha EJ, Kurz A; Crystalloid-Colloid Research Group. Hemodynamic Responses to Crystalloid and Colloid Fluid Boluses during Noncardiac Surgery. Anesthesiology. 2022 Jan 1;136(1):127-137. doi: 10.1097/ALN.0000000000004040. PMID 34724045
- [Background] Calvo-Vecino JM, Ripolles-Melchor J, Mythen MG, Casans-Frances R, Balik A, Artacho JP, Martinez-Hurtado E, Serrano Romero A, Fernandez Perez C, Asuero de Lis S; FEDORA Trial Investigators Group. Effect of goal-directed haemodynamic therapy on postoperative complications in low-moderate risk surgical patients: a multicentre randomised controlled trial (FEDORA trial). Br J Anaesth. 2018 Apr;120(4):734-744. doi: 10.1016/j.bja.2017.12.018. Epub 2018 Feb 3. PMID 29576114
- [Background] Ruetzler K, Khanna AK, Sessler DI. Myocardial Injury After Noncardiac Surgery: Preoperative, Intraoperative, and Postoperative Aspects, Implications, and Directions. Anesth Analg. 2020 Jul;131(1):173-186. doi: 10.1213/ANE.0000000000004567. PMID 31880630
- [Background] Ruetzler K, Smilowitz NR, Berger JS, Devereaux PJ, Maron BA, Newby LK, de Jesus Perez V, Sessler DI, Wijeysundera DN. Diagnosis and Management of Patients With Myocardial Injury After Noncardiac Surgery: A Scientific Statement From the American Heart Association. Circulation. 2021 Nov 9;144(19):e287-e305. doi: 10.1161/CIR.0000000000001024. Epub 2021 Oct 4. PMID 34601955
- [Background] Xu Y, Wang S, He L, Yu H, Yu H. Hydroxyethyl starch 130/0.4 for volume replacement therapy in surgical patients: a systematic review and meta-analysis of randomized controlled trials. Perioper Med (Lond). 2021 May 11;10(1):16. doi: 10.1186/s13741-021-00182-8. PMID 33971968
- [Background] Chappell D, van der Linden P, Ripolles-Melchor J, James MFM. Safety and efficacy of tetrastarches in surgery and trauma: a systematic review and meta-analysis of randomised controlled trials. Br J Anaesth. 2021 Oct;127(4):556-568. doi: 10.1016/j.bja.2021.06.040. Epub 2021 Jul 28. PMID 34330414